CLINICAL TRIAL: NCT01056159
Title: Cumulative Dose Comparison of the Efficacy and Safety of Albuterol in a Dry Powder Inhaler and an HFA MDI (Hydrofluoroalkane Metered Dose Inhaler) in Adult Patients With Asthma
Brief Title: A Cumulative Dose Study to Evaluate the Safety and Efficacy of Albuterol in a Dry Powder Inhaler and an HFA MDI (Hydrofluoroalkane Metered Dose Inhaler)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ABS-AS-101
Record Dates: First submitted 2010-01-22; First posted 2010-01-26 (Estimated); Last update posted 2022-02-02 (Actual); Status verified 2022-01

CONDITIONS: Asthma
Keywords: asthma; dry powder inhaler; short-acting beta2-agonist; SABA; bronchoconstriction; bronchodilation; bronchodilator; metered dose inhaler
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Albuterol dry powder inhaler (Experimental): The participants will receive albuterol delivered with the a DPI (dry powder inhaler) and placebo with an HFA MDI inhaler (hydrofluoroalkane metered dose inhaler).
  Interventions: Drug: Albuterol dry powder inhaler
- Albuterol HFA MDI (Active Comparator): The participants will receive albuterol delivered with an HFA MDI inhaler (hydrofluoroalkane metered dose inhaler) and placebo with albuterol in a DPI (dry powder inhaler).
  Interventions: Drug: Albuterol HFA MDI (hydrofluoroalkane metered dose inhaler)

INTERVENTIONS:
Drug: Albuterol dry powder inhaler — Albuterol DPI (dry powder inhaler) delivers 90mcg of albuterol in the excipient lactose with each inhalation. Albuterol will be given on two treatment days (3 to 14 days apart). On each treatment day albuterol will be given as a cumulative dose of 1440mcg as a series of inhalations using both Albuterol in a DPI (dry Powder inhaler) and albuterol in an HFA MDI (hydrofluoroalkane metered dose inhaler), ProAir. One inhaler will contain active drug and one inhaler will contain placebo.
  Arms: Albuterol dry powder inhaler
Drug: Albuterol HFA MDI (hydrofluoroalkane metered dose inhaler) — Albuterol HFA MDI (hydrofluoroalkane metered dose inhaler) delivers 90mcg of albuterol with each inhalation. Albuterol will be given on two treatment days (3to 14 days apart). On each treatment day albuterol will be given as a cumulative dose of 1440mcg as a series of inhalations using both Albuterol DPI (dry powder inhaler) and the comparator inhaler, albuterol HFA MDI (hydrofluoroalkane metered dose inhaler).One inhaler will contain active drug and one inhaler will contain placebo.
  Arms: Albuterol HFA MDI

SUMMARY:
The study will measure the improvement in lung function in subjects with asthma after inhaling from two inhalers, Albuterol in a dry powder inhaler and albuterol in an HFA (hydrofluoroalkane), metered dose inhaler.

DETAILED DESCRIPTION:
The study objective is to compare the efficacy and safety of albuterol in a dry powder inhaler (DPI) and albuterol in an HFA metered dose inhaler (MDI) after a cumulative dose of 1440mcg administered as 1+1+2+4+8 inhalations (90mcg per inhalation). Another study objective is to compare the pharmacokinetics (metabolism) of albuterol with the two inhalers. The pharmacokinetics of albuterol will be examined in half (24) of the study subjects. To participate in the study, patients must provide written informed consent, washout any prohibited medications and pass all the screen criteria. Once this is done, there will be two treatment visits. At each visit the subject will inhale with both types of inhalers. At each visit, one inhaler will have active drug (albuterol) and one inhaler will have placebo (dummy). The inhaler with the active drug will be switched at the two visits in a random manner. At each visit the subject will inhale with each inhaler a total of 16 times by a specific schedule. The subject will inhale from each inhaler once (1), wait 30 minutes, inhale from each inhaler once (1), wait 30 minutes, inhale from each inhaler twice (2), wait 30 minutes, inhale from each inhaler four times (4), wait 30 minutes, and then inhale from each inhaler eight times (8). The total time to complete the inhalations should be about 2 hours. Following that, there will be a series of assessments taken at regular times with vital signs measured up to 6 hours, ECG (electrocardiogram) assessed up to 4 hours, blood taken to measure potassium and glucose up to 4 hours, lung function evaluated with spirometry up to 6 hours, and for those subjects participating in the pharmacokinetic evaluation blood will be drawn up to 12 hours. The two study treatment visits will be 3 to 14 days apart. Following these visits, there will be a study concluding visit 1 to 5 days later.

ELIGIBILITY:
Inclusion Criteria:

* Must provide written informed consent,
* Must be between 18-45 years of age,
* Male or Female, females of non-child bearing potential or using reliable contraception
* Asthma for at least 6 months, FEV1 (forced expiratory volume in 1 second) between 50-80% of predicted value, and reversibility greater than or equal to 15% following 180mcg albuterol
* Stable low dose of Inhaled Corticosteroids
* Non-smoker
* Otherwise healthy
* Other criteria apply

Exclusion Criteria:

* Pregnant
* Allergic to albuterol or severe milk protein allergy
* ONLY for subject participating in PK assessments, must not have donated blood within 30 days.
* Other criteria apply

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2010-01; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Baseline-adjusted forced expiratory volume in one second (FEV1) 30 minutes after each of the five cumulative doses | At the two study treatment visits, FEV1 (forced expiratory volume in 1 second) will be measured prior to drug administration and 5 times, once at 30 minutes after each of the 5 doses.

SECONDARY OUTCOMES:
Baseline-adjusted FEV1 (forced expiratory volume in 1 second) AUC0-6 (area under the serum concentration time curve from time 0 to 6 hours) following the administration of the final cumulative dose | At the two study treatment visits, FEV1 (forced expiratory volume in 1 second) will be measured prior to drug administration and 7 time points ( 30 minutes and 1,2,3,4,5 and 6 hours) after the 5th and final dose.
ECGs (electrocardiogram) will assess the maximum and mean change from baseline of the corrected QT interval (QT interval measures the time between the start of the Q wave and the end of the T wave in the heart's electrical cycle) following study drug. | Serial ECGs (electrocardiogram) will be taken at baseline (5 minutes pre-dose), 15 minutes after each dose, and also at 30 minutes, 60 minutes, 2, 3, and 4 hours following the last cumulative dose in order to calculate the corrected QT interval.
Changes in blood pressure will be evaluated by the maximum change (systolic) and minimum change (diastolic) from baseline blood pressure, and the weighted mean change from baseline in systolic and diastolic blood pressure. | Serial measurements of systolic and diastolic blood pressure will be taken at baseline (15 minutes pre-dose), 15 minutes after each dose, and also at 30 minutes, 60 minutes, 2, 3, 4, 5, and 6 hours following the last cumulative dose.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Program Leader, Study Director — Teva Branded
Locations (8):
- United States (8):
  - Teva Clinical Study Site, Los Angeles, California
  - Teva Clinical Study Site, Denver, Colorado
  - Teva Clinical Study Site, Lakewood, Colorado
  - Teva Clinical Study Site, Normal, Illinois
  - Teva Clinical Study Site, North Dartmouth, Massachusetts
  - Teva Clinical Study Site, Minneapolis, Minnesota
  - Teva Clinical Study Site, Bellevue, Nebraska
  - Teva Clinical Study Site, Lake Oswego, Oregon